CLINICAL TRIAL: NCT04474522
Title: A Randomized Double Blind Controlled Trial of Non-invasive Preimplantation Genetic Testing for Aneuploidy and Morphology Compared With Morphology Alone in in Vitro Fertilisation
Brief Title: RCT of niPGT for Aneuploidy and Morphology Compared With Morphology Alone in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ernest Hung-Yu Ng, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: UW 20-248
Record Dates: First submitted 2020-07-06; First posted 2020-07-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Preimplantation Diagnosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group using morphology and NIPGT-A (Active Comparator): Both morphology and NIPGT-A result will be used to prioritize the sequence of embryo transfer in the intervention group.
  Interventions: Genetic: Non-invasive Preimplantation genetic testing for aneuploidy status
- control group based on morphology alone (No Intervention): Morphology only will be used to prioritize the sequence of embryo transfer in the intervention arm.

INTERVENTIONS:
Genetic: Non-invasive Preimplantation genetic testing for aneuploidy status — In the intervention group, comprehensive chromosome screening using NGS will be performed according to the recommendations of the company in all SCM samples. Sequence of replacement shall be altered by the NiPGT result after morpholgy.
  Arms: intervention group using morphology and NIPGT-A

SUMMARY:
This study is to compare the efficacy in embryo selection based on morphology alone compared to morphology and non-invasive preimplantation genetic testing for aneuploidy (NIPGT-A) in infertile women undergoing in vitro fertilization (IVF). We supposed the embryo selection based on morphology and NIPGT-A results in a higher live birth rate and a lower miscarriage rate in IVF as compared with that based on morphology alone. Therefore we would like to conduct a double-blind randomized controlled trial.

Infertile women undergoing IVF will be enrolled. The spent culture medium (SCM) of each blastocyst will be frozen individually. They will be randomized into two groups: (1) the intervention group based on morphology and NIPGT-A and (2) the control group based on morphology alone. In the control group, blastocysts with the best quality morphology will be replaced first. In the intervention group, blastocysts with the best morphology and euploid result of SCM will be replaced first.The primary outcome is a live birth per the first embryo transfer. We would like to compare live birth rates and miscarriage rates between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Women aged less than 43 years at the time of ovarian stimulation
* At least two blastocysts suitable for freezing on day 5 or 6 after oocyte retrieval

Exclusion Criteria:

* Less than two blastocysts suitable for freezing on day 5 or 6 after oocyte retrieval;
* Women undergoing PGT for monogenic diseases or structural rearrangement of chromosomes;
* Use of donor oocytes;
* Hydrosalpinx shown on pelvic scanning and not surgically treated

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 517 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Live birth | Number of live births beyond 22 weeks of gestation
  Birth beyond 22 weeks of gestation per the first FET

SECONDARY OUTCOMES:
Cumulative live birth rate | Number of pregnancies leading to live birth within 6 months of randomization
  Number of pregnancies leading to live birth within 6 months of randomization
Time to pregnancy | 1 year
  between time of IVF and pregnancy
Positive urine pregnancy test | Positive urine pregnancy test 14 days after embryo transfer
  Urine pregnancy test positive
Clinical pregnancy | 6 weeks
  Presence of intrauterine gestational sac on scanning at gestational week 6
Ongoing pregnancy | 10 weeks
  Presence of a fetal pole with pulsation at 8-10 weeks of gestation
Miscarriage defined | Pregnancy loss up to 22 weeks
  Clinically recognized pregnancy loss before the 22 weeks of pregnancy and whose denominator is the clinical pregnancy.
Multiple pregnancy | more than one intrauterine sac at 6 weeks
  presence of more than one intrauterine sac at 6 weeks of gestation
Ectopic pregnancy | 12 weeks
  Pregnancy not in the uterus
Birth weight | 1 year
  Pregnancy outcome
Apgar score | 1 year
  Pregnancy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Study Director — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spandorfer SD, Davis OK, Barmat LI, Chung PH, Rosenwaks Z. Relationship between maternal age and aneuploidy in in vitro fertilization pregnancy loss. Fertil Steril. 2004 May;81(5):1265-9. doi: 10.1016/j.fertnstert.2003.09.057. PMID 15136087
- [Background] Hassold T, Hall H, Hunt P. The origin of human aneuploidy: where we have been, where we are going. Hum Mol Genet. 2007 Oct 15;16 Spec No. 2:R203-8. doi: 10.1093/hmg/ddm243. PMID 17911163
- [Background] Nybo Andersen AM, Wohlfahrt J, Christens P, Olsen J, Melbye M. Maternal age and fetal loss: population based register linkage study. BMJ. 2000 Jun 24;320(7251):1708-12. doi: 10.1136/bmj.320.7251.1708. PMID 10864550
- [Background] Mastenbroek S, Twisk M, van der Veen F, Repping S. Preimplantation genetic screening: a systematic review and meta-analysis of RCTs. Hum Reprod Update. 2011 Jul-Aug;17(4):454-66. doi: 10.1093/humupd/dmr003. Epub 2011 Apr 29. PMID 21531751
- [Background] Yang Z, Liu J, Collins GS, Salem SA, Liu X, Lyle SS, Peck AC, Sills ES, Salem RD. Selection of single blastocysts for fresh transfer via standard morphology assessment alone and with array CGH for good prognosis IVF patients: results from a randomized pilot study. Mol Cytogenet. 2012 May 2;5(1):24. doi: 10.1186/1755-8166-5-24. PMID 22551456
- [Background] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996
- [Background] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942
- [Background] Fiorentino F, Biricik A, Bono S, Spizzichino L, Cotroneo E, Cottone G, Kokocinski F, Michel CE. Development and validation of a next-generation sequencing-based protocol for 24-chromosome aneuploidy screening of embryos. Fertil Steril. 2014 May;101(5):1375-82. doi: 10.1016/j.fertnstert.2014.01.051. Epub 2014 Mar 6. PMID 24613537
- [Background] Evans J, Hannan NJ, Edgell TA, Vollenhoven BJ, Lutjen PJ, Osianlis T, Salamonsen LA, Rombauts LJ. Fresh versus frozen embryo transfer: backing clinical decisions with scientific and clinical evidence. Hum Reprod Update. 2014 Nov-Dec;20(6):808-21. doi: 10.1093/humupd/dmu027. Epub 2014 Jun 10. PMID 24916455
- [Background] Lee E, Illingworth P, Wilton L, Chambers GM. The clinical effectiveness of preimplantation genetic diagnosis for aneuploidy in all 24 chromosomes (PGD-A): systematic review. Hum Reprod. 2015 Feb;30(2):473-83. doi: 10.1093/humrep/deu303. Epub 2014 Nov 28. PMID 25432917
- [Background] Munne S, Kaplan B, Frattarelli JL, Child T, Nakhuda G, Shamma FN, Silverberg K, Kalista T, Handyside AH, Katz-Jaffe M, Wells D, Gordon T, Stock-Myer S, Willman S; STAR Study Group. Preimplantation genetic testing for aneuploidy versus morphology as selection criteria for single frozen-thawed embryo transfer in good-prognosis patients: a multicenter randomized clinical trial. Fertil Steril. 2019 Dec;112(6):1071-1079.e7. doi: 10.1016/j.fertnstert.2019.07.1346. Epub 2019 Sep 21. PMID 31551155
- [Derived] Cheng HYH, Chow JFC, Lam KKW, Lai SF, Yeung WSB, Ng EHY. Randomised double-blind controlled trial of non-invasive preimplantation genetic testing for aneuploidy in in vitro fertilisation: a protocol paper. BMJ Open. 2023 Jul 27;13(7):e072557. doi: 10.1136/bmjopen-2023-072557. PMID 37500277